CLINICAL TRIAL: NCT04250571
Title: Taking Open Label Placebo Further: Randomized Controlled Trial of Imaginary Pills in Test Anxiety
Brief Title: Taking Open Label Placebo Further: Trial of Imaginary Pills in Test Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Prof. Dr., Jens Gaab, Division of Clinical Psychology and Psychotherapy, University of Basel, Switzerland (Unknown); Emer. Prof. Dr., Irving Kirsch, Universities of Hull and Plymouth, United Kingdom, and University of Connecticut, USA (Unknown); Cand. psych., Niels Bagge, Institut for Emotionsfokuseret Terapi, Roskilde, Denmark (Unknown); Asst. Prof. Dr., Claudia Carvalho, Department of Clinical and Health Psychology ISPA, Lisbon, Portugal (Unknown); Dr. phil., Cosima Locher, Boston Children's Hospital, Harvard Medical School, Boston, MA, USA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 035-19-1; ex20Gaab
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Test Anxiety
Keywords: imaginary pills; open label placebo (OLP) treatment; placebo
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No treatment group (Experimental): Participants will receive no pills and will be told that they are in the no treatment group
  Interventions: Other: information about "No treatment group"
- Imaginary pill (IP) group (Experimental): Participants will be instructed to take an imagined pill. This instruction consists of a procedure including five steps (i.e., identifying the IP sensitive problem, building trust/belief/reality of the IP, constructing a personally meaningful IP, taking the IP, suggestions for self-administering the IP in real life, and building adherence)
  Interventions: Other: imaginary pill technique
- Open label placebo group (Experimental): Participants will have the information that they are receiving inert pills (i.e. "P-Dragees", containing "Placebo")
  Interventions: Other: open label placebo

INTERVENTIONS:
Other: information about "No treatment group" — Participants will receive no pills and will be told that they are in the no treatment group
  Arms: No treatment group
Other: imaginary pill technique — Participants will be instructed to take an imagined pill. This instruction consists of a procedure including five steps (i.e., identifying the IP sensitive problem, building trust/belief/reality of the IP, constructing a personally meaningful IP, taking the IP, suggestions for self-administering the IP in real life, and building adherence). Participants in this group receive daily e-mail reminders.
  Arms: Imaginary pill (IP) group
Other: open label placebo — Participants will have the information that they are receiving inert pills (i.e. "P-Dragees", containing "Placebo"), combined with the following scientific rationale: (a) deceptive as well as open label placebos have been found to be effective in relieving symptoms in a variety of clinical conditions namely anxiety, depression, chronic pain (the placebo effect is powerful), (b) classical conditioning are one of the possible mechanism of this effect (the body automatically responds), (c) positive expectations may help but are not necessary, (suspend disbelief), (d) compliance with these instructions are important for outcome (taking the pills faithfully is important).
  Participants in this group receive daily e-mail reminders.
  Arms: Open label placebo group

SUMMARY:
Employing imaginary pills could offer a new way of investigating underlying mechanisms of open label placebo (OLP) treatment by eliminating the physical treatment constituent (i.e., the pill itself). This can reveal the power of the purely psychological component of a placebo and gives insights into underlying mechanisms of placebo effects. The aim of the project is to assess possible effects of an imaginary pill in comparison to no treatment, and open label placebo treatment in subjects with test anxiety.

Interventions (seven to three weeks before the exam) will be held online using a video Chat application such as zoom (https://zoom.us/) or skype (https://www.skype.com/de/) or will take place at the division of Clinical Psychology and Psychotherapy, University of Basel (Missionsstrasse 62, 4055 Basel).

ELIGIBILITY:
Inclusion Criteria:

* Having an exam at the end of the semester, that is still at least four weeks ahead
* Self-reported fear of the exam (i.e., not clinical)
* Healthy by self-report statement (i.e., no known current or chronic somatic diseases or psychiatric disorders)
* Willing to participate in study

Exclusion Criteria:

* Any acute or chronic disease (chronic pain, hypertension, heart disease, renal disease, liver disease, diabetes)
* Current medications (psychoactive medication, narcotics, intake of analgesics)
* Any psychiatric disorders or being currently in psychological or psychiatric treatment
* Insufficient German language skills to understand the instructions
* Daily consumption of more than three alcoholic standard beverages (a standard alcoholic beverage is defined as either 3dl beer or 1 dl wine or 2cl spirits)
* Current or regular drug consumption
* Being a master student in Psychology
* Allergy of one of the ingredients of the placebo pills (P-Dragees blue Lichtenstein)
* Problems to swallow pills

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Prüfungsangstfragebogen (PAF) questionnaire | from seven to three weeks before the exam (t0; baseline assessment), after study visit (t1) once a week for the following two weeks (t2-t3; midpoint assessments), baseline (t0 = 4 weeks to exam)) to posttreatment (t4 = 2to 0 days to exam )
  The PAF questionnaire consisting of 20 items with four subscales (worry, emotionality, interference, lack of confidence) is a multi-faceted measure of test anxiety. Each subscale consists of five items with a total of 20 questions overall. Response on a 4-point Likert-scale ranging from 1 (almost never) to 4 (almost always).

SECONDARY OUTCOMES:
Change in the Pittsburgh Sleep Quality Index (PSQI) | from seven to three weeks before the exam (t0; baseline assessment), after study visit (t1) once a week for the following two weeks (t2-t3; midpoint assessments), baseline (t0 = 4 weeks to exam)) to posttreatment (t4 = 2to 0 days to exam )
  The PSQI is an 18 item self-rating questionnaire forming 7 subscales and includes frequency of sleep disturbing events, the assessment of sleep quality, the usual sleep times, sleep latency and sleep duration, the intake of sleep medications, as well as daytime fatigue.
Change in Change-sensitive symptom list (ASS-SYM symptom list) | from seven to three weeks before the exam (t0; baseline assessment), after study visit (t1) once a week for the following two weeks (t2-t3; midpoint assessments), baseline (t0 = 4 weeks to exam)) to posttreatment (t4 = 2to 0 days to exam )
  ASS-SYM symptom list It is composed of 48 items arranged in 6 subscales: physical and psychological exhaustion, nervousness and mental tension, psycho-physiological dysregulation, performance and behavioral problems, burden of pain as well as self-determination and self-control problems.
test performance | assessed two months after the exam
  test performance (i.e., grade of the respective exam or pass/fail) of each participant
semi-structured qualitative interview with open-ended questions | 30-60 min duration after personal study conclusion (1 to 5 weeks after exam)
  qualitative interview to assess the subjective experiences, opinions and perceptions of (1) receiving the imaginary pill (N=10) and open label placebo (N=10) treatment, (2) their experiences during the three week intervention phase, (3) the exam situation (4) and thoughts about the use in the future. Participants of the no treatment group are not included. The data will be analyzed using a qualitative content analysis after Mayring (Mayring, 2014)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Buergler, M. Sc., Principal Investigator — Division of Clinical Psychology and Psychotherapy, University of Basel
Locations (1):
- Division of Clinical Psychology and Psychotherapy, Department of Psychology, University of Basel, Basel, Switzerland

REFERENCES:
- [Background] Buergler S, Sezer D, Bagge N, Kirsch I, Locher C, Carvalho C, Gaab J. Imaginary pills and open-label placebos can reduce test anxiety by means of placebo mechanisms. Sci Rep. 2023 Feb 14;13(1):2624. doi: 10.1038/s41598-023-29624-7. PMID 36788309